CLINICAL TRIAL: NCT01340170
Title: An Open, Non-randomized, Prospective Multi-centre Study Evaluating a Soft Bone Drilling Protocol for Single Tooth Restoration in the Posterior Area With Immediate Loading
Brief Title: A Study Evaluating OsseoSpeed TX Using Different Drilling Protocols With Immediate Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-OTX-0002
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-03

CONDITIONS: Edentulism

ARMS (2):
- Soft bone drilling protocol (Experimental): A soft bone drilling protocol will be used in bone quality 3 and 4
  Interventions: Device: OsseoSpeed TX
- Standard drilling protocol (Active Comparator): A standard drilling protocol will be used in bone quality 1 and 2
  Interventions: Device: OsseoSpeed TX

INTERVENTIONS:
Device: OsseoSpeed TX — OsseoSpeed TX dental implants, 6-17 mm

SUMMARY:
This study is initiated to support the OsseoSpeedTM TX implant with clinical data showing that a soft bone drilling protocol and immediate loading does not have any important negative effect on marginal bone level maintenance.

DETAILED DESCRIPTION:
This study is designed to evaluate a soft bone drilling protocol compared to a standard bone drilling protocol when using OsseoSpeedTM TX with regards to marginal bone level changes and implant survival rate one year after loading. The aim is also to investigate potential differences in initial stability and in general user friendliness between the two drilling protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Female/male aged 18 years and over
3. History of edentulism in the study area of at least 3 months
4. At least 4 months healing after last grafting procedure in the study area
5. In need for implant treatment replacing one to four missing single tooth in positions 14-17, 24-27, 34-37 and 44-47
6. The study implant position must be surrounded by natural tooth roots, unless the implant will constitute the most distal dentition.
7. Deemed by the investigator to be suitable for one stage surgery
8. Deemed by the investigator to be suitable for immediate loading
9. Deemed by the investigator as likely to present an initially stable implant situation.
10. Deemed by the investigator to have a "functional" opposing dentition at the time of loading the implants.

Exclusion Criteria

1. Unlikely to be able to comply with study procedures, as judged by the investigator
2. Uncontrolled pathological processes in the oral cavity
3. Known or suspected current malignancy
4. History of radiation therapy in the head and neck region
5. History of chemotherapy within 5 years prior to surgery
6. Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
7. Uncontrolled diabetes mellitus
8. Corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
9. Present alcohol and/or drug abuse
10. Current need for bone grafting and/or augmentation in the planned implant area
11. Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
12. Previous enrolment in the present study.
13. Simultaneous participation in another clinical study, or participation in a clinical study during the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruggero Rodriguez y Baena, Prof, Principal Investigator — University of Pavia
Locations (9):
- Italy (9):
  - Studio Associato Maffei, Bari
  - Studio Dentistico Paolo Torrisi, Catania
  - Societa diMedicina Odontostomatologica Srl, Como
  - Dept. of Oral Sciences "S. Palazzi", University of Pavia, Pavia
  - Studio Dentistico, Perugia
  - La Scala & Partners Studio Associato, Pistoia
  - Studio Odontoiatrico, Roma
  - Studio Dentistico, Torino
  - Studio Polispecialistico di Odontoiatria, Udine

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Groups:
- Standard Drilling Protocol (Group A): A standard drilling protocol will be used in bone quality 1 and 2
  OsseoSpeed TX: OsseoSpeed TX dental implants, 6-17 mm
- Soft Bone Drilling Protocol (Group B): A soft bone drilling protocol will be used in bone quality 3 and 4
  OsseoSpeed TX: OsseoSpeed TX dental implants, 6-17 mm
- Group A + B: Subjects with implants from both Group A and Group B
Period: Overall Study
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B) | Group A + B
Started (ITT population) | 79; 83 Implants | 86; 99 Implants | 3; 6 Implants (Three participants received six implant treatments defined as Group A (3 implants) and Group B (3 implants) respectively. These implants are not included in "Group A" and "Group B", but instead in Group "A + B". Outcome measure 1 to 8 are analyzed on implant level only and do not contain subject level group "Group A + B".)
Permanent Restoration (Start + 3 Months) (ITT population) | 79; 83 Implants | 81; 94 Implants | 3; 6 Implants (Three participants received six implant treatments defined as Group A (3 implants) and Group B (3 implants) respectively. These implants are not included in "Group A" and "Group B", but instead in Group "A + B". Outcome measure 1 to 8 are analyzed on implant level only and do not contain subject level group "Group A + B".)
Completed (ITT population) | 76; 79 Implants | 79; 91 Implants | 3; 6 Implants (Three participants received six implant treatments defined as Group A (3 implants) and Group B (3 implants) respectively. These implants are not included in "Group A" and "Group B", but instead in Group "A + B". Outcome measure 1 to 8 are analyzed on implant level only and do not contain subject level group "Group A + B".)
Not Completed | 3; 4 Implants | 7; 8 Implants | 0; 0 Implants
Not completed — Lost to Follow-up | 2 | 4 | 0
Not completed — Implant failure | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B) | Group A + B | Total
Number analyzed (Participants) | 79 | 86 | 3 | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (12.6) | 47.5 (12.3) | 54.3 (17.7) | 47.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 3 | 90
  Male | 36 | 42 | 0 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Level Change
Description: Marginal Bone Level alterations will be determined from radiographs and expressed as the difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant.
Time Frame: Implant insertion and 12 months post implant insertion
Population: ITT subjects with MBL data available (MBL data missing for 14 implants in Group A, and from 10 implants in group B). Outcome measure 1 is analyzed on implant level only and does not contain subject level group "Group A + B".
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B)
Number analyzed (Participants) | 63 | 72
Number analyzed (Implants) | 68 | 84
mm | -0.25 (0.9) | -0.2 (0.67)

2. Secondary Outcome: Marginal Bone Level Change
Description: as for outcome 1
Time Frame: Implant insertion and 3 months post implant insertion
Population: ITT subjects with MBL data available (MBL data missing from 10 implants in Group A, from 9 implants in group B). Outcome measure 2 is analyzed on implant level only and does not contain subject level group "Group A + B".
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B)
Number analyzed (Participants) | 71 | 75
Number analyzed (Implants) | 76 | 88
mm | -0.2 (0.62) | -0.29 (0.67)

3. Secondary Outcome: Implant Survival Rate
Description: Implant survival rate will be evaluated by both clinically and radiographically counting the number of remaining implants from implant placement to one year after loading.
Time Frame: 12 months after baseline, i.e., implant insertion
Population: ITT subjects at 12 months as well as known implant failures already terminated are included in the analysis.
  Outcome measure 3 is analyzed on implant level only and does not contain subject level group "Group A + B".
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B)
Number analyzed (Participants) | 77 | 83
Number analyzed (Implants) | 84 | 98
Implants
  Implants confirmed success | 82 | 94
  Implants confirmed failure | 2 | 4

4. Secondary Outcome: Implant Stability Assessed Clinically/Manually
Description: Evaluated clinically/manually and recorded as stable yes/no.
Time Frame: At implant insertion
Population: ITT population. Outcome measure 4 is analyzed on implant level only and does not contain subject level group "Group A + B".
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B)
Number analyzed (Participants) | 79 | 86
Number analyzed (Implants) | 86 | 102
Implants
  Implant stability - Yes | 86 | 97
  Implant stability - No | 0 | 5

5. Secondary Outcome: Implant Stability Using Resonance Frequency Analysis (RFA)
Description: The Osstell® instrument "Osstell® ISQ" will be used to measure RFA. RFA measures the frequency with which a device vibrates. By comparing resonance frequencies the stability of a dental implant can be determined as the resonance frequency changes with different stability. The Osstell® ISQ instrument translates the RFA value into an Implant Stability Quotient (ISQ) scale value. ISQ is a scale from 1 to 100. The ISQ scale has a non-linear correlation to micro mobility, with a higher value corresponding to increased stability.
Time Frame: At implant insertion.
Population: ITT population. Outcome measure 5 is analyzed on implant level only and does not contain subject level group "Group A + B".
Measure: Mean (Standard Deviation); unit: ISQ on implant level
Units Other Than Participants: Implants
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B)
Number analyzed (Participants) | 79 | 86
Number analyzed (Implants) | 86 | 102
ISQ on implant level
  Mesio-Distal | 78.6 (6.2) | 77.5 (9.6)
  Bucco-Palatinal | 78.8 (5.9) | 77.7 (9.4)

6. Secondary Outcome: Perception During Implant Insertion - "The Implant Was Guided Into the Prepared Osteotomy"
Description: After implant insertion, a questionnaire will be completed for each study implant by the surgeon. The questionnaire contains following statements "The implant was guided into the prepared osteotomy", "The implant followed the prepared osteotomy" and "The implant has a good primary stability". The surgeon records his/her response to each statement with a number from 1 to 10 , where 1= totally disagree with the statement, and 10= totally agree with the statement.
Time Frame: After implant insertion
Population: ITT subjects. Outcome measure 6 is analyzed on implant level only and does not contain subject level group "Group A + B".
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B)
Number analyzed (Participants) | 79 | 86
Number analyzed (Implants) | 86 | 102
score on a scale | 7.5 (2.6) | 7.1 (2.4)

7. Secondary Outcome: Perception During Implant Insertion - "The Implant Followed the Prepared Osteotomy"
Description: as for outcome 6
Time Frame: After implant insertion
Population: ITT subjects. Outcome measure 7 is analyzed on implant level only and does not contain subject level group "Group A + B".
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: implants
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B)
Number analyzed (Participants) | 79 | 86
Number analyzed (implants) | 86 | 102
score on a scale | 8.2 (1.6) | 7.6 (2.0)

8. Secondary Outcome: Perception During Implant Insertion - "The Implant Has a Good Primary Stability"
Description: as for outcome 6
Time Frame: After implant insertion
Population: ITT subjects. Outcome measure 8 is analyzed on implant level only and does not contain subject level group "Group A + B".
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: implants
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B)
Number analyzed (Participants) | 79 | 86
Number analyzed (implants) | 86 | 102
score on a scale | 8.7 (1.3) | 8.1 (1.7)

ADVERSE EVENTS:
Time Frame: From enrollment up to study termination, i.e., 1 year post implant insertion.
Arm/Group | Standard Drilling Protocol (Group A) | Soft Bone Drilling Protocol (Group B) | Group A + B
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/86 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/86 | 0/3
Other Adverse Events (participants affected / at risk) | 0/79 | 0/86 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No